CLINICAL TRIAL: NCT06226636
Title: Diagnostic Accuracy of Using an Immediate Pressor Response to Oral Salt (IPROS) to Identify Salt Sensitivity of Blood Pressure (SSBP): a Time Series Clinical Trial
Brief Title: Immediate Pressor Response to Oral Salt
Acronym: IPROS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mulungushi University (Other)
Responsible Party: Principal Investigator, Sepiso K. Masenga, Senior Lecturer, Mulungushi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IPROS
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): intervention given
  Interventions: Other: salt

INTERVENTIONS:
Other: salt — After ≥8 hr overnight fasting, participants will be required to ingest 780 mg of sodium (2 g salt) and BP measured every 10 minutes for 2 hours to determine IPROS. For SSBP, Participants are put on low salt (50 mmol Na/day) followed by seven days of high salt diet (250 mmol Na/day). Participants' mean arterial pressure (MAP) difference between low- and high-salt diet will be used to define salt sensitivity (MAP≥8 mmHg) and salt resistance (MAP≤5 mmHg).

SUMMARY:
The goal of this study is to establish a diagnostic accuracy of an immediate pressor response to oral salt (IPROS) to identify salt sensitivity of blood pressure (SSBP)

DETAILED DESCRIPTION:
Participants are given dietary salt and their BP is measured every 10 minutes for 2 hours. IPROS is diagnosed with significant mean arterial pressure increase

For SSBP, participants are put on high salt diet for a week and monitored and low salt week. The Mean arterial pressure difference between high salt and low salt is used to diagnose SSBP

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are males or females, aged 18-65 years.

Exclusion Criteria:

* Kidney disease, Cardiovascular disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
SSBP | 2 weeks
  Salt sensitivity status

SECONDARY OUTCOMES:
IPROS | 2 hours
  Immediate pressor response

CONTACTS AND LOCATIONS:
Locations (2):
- Zambia (2):
  - Livingstone University Teaching Hospital, Livingstone, Southern Province
  - Kanyama General Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Data set and manuscripts published
Supporting Information: CSR
Time Frame: 2025
Access Criteria: email